CLINICAL TRIAL: NCT05287022
Title: Use of Nasal Nitric Oxide Testing in Improving Primary Ciliary Dyskinesia Clinical Care
Status: Recruiting | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 260432
Record Dates: First submitted 2021-04-09; First posted 2022-03-18 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Primary Ciliary Dyskinesia
Keywords: nNO; Diagnosis; PCD
MeSH Terms: conditions — Ciliary Motility Disorders; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
this study is aiming at learning more about primary ciliary dyskinesia (PCD) and tests that are used to diagnose this condition. One purpose of this study is to measure the level of nitric oxide in the nasal passages and examine how often the results correlate with other tests currently done to make the diagnosis.

DETAILED DESCRIPTION:
This will be an observational study. Participants who are referred by their clinician for nasal NO testing and meet the inclusion and exclusion criteria will be allowed to undergo testing. Informed consent will be completed prior to testing. The participant and/or guardian will be informed that this testing is not a clinically approved test at this time and thus it cannot confirm diagnosis of PCD. This test is to correlate with other diagnostic tests so that in the future it can be an approved diagnostic test. Data will be collected from the electronic medical records regarding participants.

The data collected will be stored on a REDCap (Research Electronic Data Capture) registry. The registry will contain participants' direct identifiers (like medical record). De-identified data will be used from the registry for monitoring, further analysis and presentations. The results of the testing may be included in the medical chart of each participant as part of the diagnosis discussion with family.

Consent forms will be obtained from participants >18 years of age or who are emancipated minors, or guardian for patients <18 years of age. Guardian refers to parent, guardian, or legally authorized personnel throughout this document.

The data collected will be used to refine and improve the diagnostic testing for PCD at Arkansas Children's Hospital. This will also involve collaboration with other sub-specialties like otolaryngology and allergy/immunology. With continued research regarding nasal nitric oxide testing, this may involve the use of this test as a screening tool for PCD in the right clinical setting. This will involve analyzing the association of nasal nitric oxide levels with approved diagnostic tests (ciliary biopsy and genetic testing).

Testing will be completed using (Eco-Physics Analyzer CLD 88 sp with DENOX 88). this testing will be done in the Arkansas Children's hospital pulmonary function laboratory, once all training is completed.

This equipment is not currently FDA approved for PCD diagnostic testing and therefore, referring clinicians will be informed of the results of this test and its limitations as a research tool will be discussed. However, there is growing evidence that this testing has utility as a non-invasive screening tool for PCD and continued data from the general pediatric pulmonary population is needed.

In addition to being non-invasive testing, it has very little risk as it simply monitors nasal nitric oxide levels in the sinus cavities during regular breathing without sedation. There is ongoing research to better determine normative values and thresholds for further PCD confirmatory testing, especially in the younger population. In the general population this testing has a greater negative predictive value than a positive predictive value. Consequently, the testing will be done on individuals who have at least two of the following clinical criteria for PCD: history of neonatal respiratory distress, chronic rhinitis, chronic cough, or situs defects.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are diagnosed with Primary Ciliary Dyskinesia OR
* Individuals with abnormal PCD diagnostics (abnormal ciliary biopsy or PCD genetics) OR
* Individuals with unexplained bronchiectasis OR
* Individuals undergoing PCD diagnostic testing (ciliary biopsy, PCD genetic testing) or concern based on clinical symptoms (at least two of the following):

  * Neonatal respiratory distress
  * Organ laterality defects
  * Year-round cough starting in first year of life or bronchiectasis on chest CT
  * Year-round nasal congestion starting in first year of life or pansinusitis
  * Multiple ear infections in the first two years of life with sequelae (e.g. ear tubes, chronic effusion, abnormal audiological exam)
  * History of recurrent pneumonias (at least 2 in one year or more than 3 at any time)
* Ability to provide consent for participation in study by the participants or guardian
* Ability to perform the test
* Age >= 2 years of age

Exclusion Criteria:

* Individuals who are unable to understand the requirements of the study.
* Individuals (or guardians) who are unwilling to provide consent.
* Individuals who are unable to complete the testing
* Recent history of sinus surgery (within four weeks) or bloody nose (within one week) of testing (they can be included at a later date)
* Patients who are currently being treated (within one week) with antibiotics for sinusitis or respiratory symptoms (they can be included at a later date)
* Age <2 years of age

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will include individuals who are diagnosed with PCD or undergoing work-up for primary ciliary dyskinesia based on their clinical symptoms as determined by the primary pulmonologist or other specialist
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Measuring nasal nitric oxide in comparison to ciliary biopsy and genetic testing for the diagnosis of PCD | throughout the study, an average of 3 years
  Individuals with PCD have characteristically low values of nNO; values below an established cut-off of 77nL/min are strongly associated with PCD in compatible clinical settings. These values are not well established for individuals who are in 2-5 years of age. nNO measurements (in nL/min) in 2-5 years of age will be compared to the diagnosis of PCD and assessed to establish diagnostic cut-offs.

SECONDARY OUTCOMES:
Comparing tidal breathing to resistor method | throughout the study, an average of 3 years
  comparing nNO values in nL/min obtained via tidal breathing technique to those obtained via resistor method.

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

REFERENCES:
- [Background] Shapiro AJ, Davis SD, Polineni D, Manion M, Rosenfeld M, Dell SD, Chilvers MA, Ferkol TW, Zariwala MA, Sagel SD, Josephson M, Morgan L, Yilmaz O, Olivier KN, Milla C, Pittman JE, Daniels MLA, Jones MH, Janahi IA, Ware SM, Daniel SJ, Cooper ML, Nogee LM, Anton B, Eastvold T, Ehrne L, Guadagno E, Knowles MR, Leigh MW, Lavergne V; American Thoracic Society Assembly on Pediatrics. Diagnosis of Primary Ciliary Dyskinesia. An Official American Thoracic Society Clinical Practice Guideline. Am J Respir Crit Care Med. 2018 Jun 15;197(12):e24-e39. doi: 10.1164/rccm.201805-0819ST. PMID 29905515
- [Background] Shapiro AJ, Zariwala MA, Ferkol T, Davis SD, Sagel SD, Dell SD, Rosenfeld M, Olivier KN, Milla C, Daniel SJ, Kimple AJ, Manion M, Knowles MR, Leigh MW; Genetic Disorders of Mucociliary Clearance Consortium. Diagnosis, monitoring, and treatment of primary ciliary dyskinesia: PCD foundation consensus recommendations based on state of the art review. Pediatr Pulmonol. 2016 Feb;51(2):115-32. doi: 10.1002/ppul.23304. Epub 2015 Sep 29. PMID 26418604
- [Background] Shapiro AJ, Dell SD, Gaston B, O'Connor M, Marozkina N, Manion M, Hazucha MJ, Leigh MW. Nasal Nitric Oxide Measurement in Primary Ciliary Dyskinesia. A Technical Paper on Standardized Testing Protocols. Ann Am Thorac Soc. 2020 Feb;17(2):e1-e12. doi: 10.1513/AnnalsATS.201904-347OT. PMID 31770003
- [Background] Collins SA, Behan L, Harris A, Gove K, Lucas JS. The dangers of widespread nitric oxide screening for primary ciliary dyskinesia. Thorax. 2016 Jun;71(6):560-1. doi: 10.1136/thoraxjnl-2015-208056. Epub 2016 Feb 19. PMID 26896442